CLINICAL TRIAL: NCT02962908
Title: A Randomised, Double-blind, Placebo-controlled, Single-centre Phase IIb Trial as Part of the EU-funded UNISEC Project to Assess the Immunogenicity and Safety of Different Formulations and Dosing Regimens of FLU-v Vaccine in Healthy Adults
Brief Title: A Randomised, Double-blind, Placebo-controlled Phase IIb Trial to Test FLU-v Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTcell Limited (Industry)
Collaborators: Seventh Framework Programme (Other); University of Groningen (Other); University Medical Center Groningen (Other); Robert Koch Institut (Other Government); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU-v 003; 2015-001932-38 (EudraCT Number)
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Influenza
Keywords: broad; universal; vaccine; influenza; peptide; Tcell; UNISEC
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): (n=74): FLU-v on Day 0 and Day 21
  Interventions: Biological: FLU-v
- Group 2 (Experimental): (n=74): adjuvanted FLU-v on Day 0, saline (0.5mL) on Day 21
  Interventions: Biological: adjuvanted FLU-v; Biological: Saline
- Group 3 (Placebo Comparator): (n=37): saline solution (0.5ml) on Day 0 and Day 21
  Interventions: Biological: Saline
- Group 4 (Placebo Comparator): (n=37): Adjuvanted placebo on Day 0, saline (0.5mL) on Day 21
  Interventions: Biological: Saline; Biological: Adjuvanted placebo

INTERVENTIONS:
Biological: FLU-v — Subcutaneous injection in the upper arm with 500 ug of FLU-v as 0.5ml suspension in 0.01M HCl and 0.01M NaOH
  Arms: Group 1
Biological: adjuvanted FLU-v — Subcutaneous injection in the upper arm with 500ug of FLU-v emulsified in 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection
  Arms: Group 2
Biological: Saline — Subcutaneous injection in the upper arm with 0.5ml of saline
  Other Names: NaCl
  Arms: Group 2; Group 3; Group 4
Biological: Adjuvanted placebo — Subcutaneous injection in the upper arm with an emulsion made with 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection
  Arms: Group 4

SUMMARY:
FLU-v is a vaccine that aims to protect against a wide range of flu viruses. The purpose of this study is to measure the immune responses induced by FLU-v vaccine. This study will look at how safe FLU-v is when administered and how successful it is in preventing flu or reducing the severity of the flu symptoms.

The study requires 222 healthy volunteers 18-60 years old. Participation in the study will take a maximum of 7 months and consists of 5 visits. During visit 1, subjects will be examined by a doctor to make sure they are eligible to enter the study. A 15ml blood sample (a tablespoon) will be taken to check general health followed by a general physical exam. Medical history and some personal information will be collected. Subjects that have received the traditional flu vaccine in the past 6 months, and those females who are pregnant or breastfeeding will not be allowed in the study. Subjects of childbearing age must agree to use effective contraceptive methods.

At visit 2, subjects will be randomly allocated to one of the four treatment groups summarised below:

* Treatment 1: FLU-v (test vaccine) at the start of the study (Day 0) and then again 21 days later
* Treatment 2: FLU-v (test vaccine) with an additional substance added [known as Montanide ISA 51] which improves the effect of the test vaccine. Injection will be given on Day 0 and then Placebo (no test vaccine) alone 21 days later
* Treatment 3: Placebo (no test vaccine) injection on Day 0 and then 21 days later
* Treatment 4: Placebo (no test vaccine) with an additional substance added [known as Montanide ISA 51] on Day 0 and then Placebo (no test vaccine) alone 21 days later Treatment will be injected under the skin in the upper arm on day 0 (visit 2) and 21 days later (visit 3). Blood samples will be taken before treatment (day 0), and on days 42 (visit 4) and 180 (visit 5) to the immune responses induced by the vaccine.

Subjects will be asked to complete a diary card to write down any side effects that they may experience after vaccination. Subjects will also be asked to complete another diary card to document any flu-like symptoms experienced between December 2016 and March 2017, this time is officially considered as the flu season. During this period, if the subject experiences flu-like symptoms, a collection of a nose and tonsil swab will be arranged by the study site to confirm whether they have the flu or not.

DETAILED DESCRIPTION:
Rationale: Current seasonal influenza vaccines mainly induce immune responses against viral membrane glycoproteins. These proteins, however, undergo continuous mutations by a process called antigenic drift. To prevent immune escape, annual vaccination with the latest predicted viral strains is adopted. Such vaccination strategy not only poses inconvenience and cost-inefficiency, but also results in poor protective effectiveness when the vaccinated strains are mismatched with the actual circulating strains. The latter point is especially of concern during a pandemic outbreak, when a large geographical area is affected and the general population is naïve to the newly re-assorted viral strain due to antigenic shift.

Objective: To evaluate the safety and immunogenicity of the influenza vaccine (FLU-v, as a suspension or adjuvanted as emulsion) targeting conserved immunogenic regions of influenza A and B viruses in healthy adults, in particular to show that the TH1 cytokine response at 42 and 180 days after the first injection is greater in the adjuvanted FLU-v and unadjuvanted FLU-v than in the placebo.

Study design: A total of 222 study participants will be recruited. The study follows a factorial design where the two factors are treatment (FLU-v / placebo) and formulation (unadjuvanted / suspension, adjuvanted / emulsion). Subjects will be randomised in two strata (age 18 to 40, age 41 to 60) to one of the following treatment regimens:

* Group 1 (n=74): FLU-v (unadjuvanted) as a suspension in pH neutral HCl/NaOH (0.5mL) on Day 0 and Day 21
* Group 2 (n=74): (0.5mL) ISA-51-adjuvanted FLU-v emulsified in water for injection (WFI) on Day 0, saline (0.5mL) on Day 21
* Group 3 (n=37): saline solution (0.5mL ) on Day 0 and Day 21
* Group 4 (n=37): WFI and ISA-51 emulsion (0.5mL) on Day 0, saline (0.5mL) on Day 21

Each administration will be given subcutaneously. Solicited and unsolicited adverse events (AEs) will be collected by AE questionnaire/diary card until day 42. Adverse events (AEs) and serious adverse events (SAEs) will be collected for the entire study period. The treatments will be administered starting in third quarter of 2016 in order to provide protection for the subsequent influenza season starting in December 2016. Blood samples will be taken from all subjects on day 0 (before FLU-v vaccination), 42 (21 days after the second dosing) and 180 (159 days after the second dosing) for the evaluation of FLU-v-specific cellular and humoral immune responses. Clinical symptom scores to ascertain severity and the incidence of RT-PCR-confirmed influenza A and/or B infection will be recorded during the subsequent influenza season (December 2016 to March 2017) to decide clinical efficacy of the tested vaccines.

Study population: Healthy volunteers aged 18-60 years. Intervention: FLU-v investigational influenza vaccine lyophilised product containing 500 micrograms of total peptides reconstituted in either 0.01M HCl (0.25ml) and 0.01M NaOH (0.25ml) to achieve a volume of 0.5ml, or emulsified in WFI (water for injection, 0.25ml) and ISA-51 (0.25ml) to achieve a volume of 0.5ml.

Primary study parameters/endpoints: For immunogenicity: To compare the change from baseline (Day 0) between treatments in cellular immune responses, specifically TH1 cytokines, in all groups 42 and 180 days following FLU-v vaccination. For safety: (1) To evaluate the solicited AEs in all subjects until 21 days after the last dosing of the study vaccine (FLU-v); (2) To evaluate the unsolicited AEs and SAEs in all subjects for the entire study period after the first dosing of FLU-v.

Secondary study parameters/endpoints: To evaluate the humoral immune responses specific to FLU-v and TH2 cytokines from baseline in all groups 42 and 180 days following FLU-v vaccination.

Exploratory study parameters/endpoints: For immunogenicity: To evaluate the change from baseline in cellular immune responses based on additional CMI assays such as ELISPOT (Enzyme-Linked ImmunoSpot) in all groups at 42 and 180 days following FLU-v vaccination, in a subset of subjects chosen at random.

Clinical efficacy: (1) To evaluate the efficacy of FLU-v vaccine in reducing the incidence of RT-PCR confirmed influenza A and/or B infections in all subjects during the influenza season 2016-2017. (2) To evaluate the efficacy of FLU-v vaccine in the reduction of symptom score among RT-PCR confirmed influenza A and/or B infection cases during the influenza season 2016-2017. The relationship between efficacy and cellular and humoral response will be explored if possible.

The effect of previous influenza vaccination on the immunogenicity of FLU-v will be assessed in a post-hoc exploratory analysis after stratification of the data based on exposure to the influenza vaccine in the previous 24 months or over.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The intended application of the IMP is as a prophylactic vaccine to prevent influenza virus infection by inducing an enhanced influenza-specific immune response. The FLU-v vaccine is designed to be delivered either as a naturally particulate suspension (i.e. no adjuvant) or emulsified in adjuvant. Particulate and emulsified protein preparations are preferentially taken up by phagocytic cells (e.g. dendritic cells) responsible for inducing primary immune responses.

Treatment with FLU-v of up to four doses of 263 μg/occasion or up to two doses of 553 μg/occasion, with or without adjuvant, was well tolerated in animals with no signs of systemic toxicity. In pre-clinical studies, subcutaneous administration of ISA 51 resulted in no systemic toxicity. At the injection sites and occasionally in adjacent tissue the injected material remained surrounded by a mild chronic inflammatory response. As the IMP is provided in one presentation (500 μg of the combined peptide) in lyophilized form for suspension in a sealed single-use vial, overdose is highly unlikely.

In a single centre, randomised, double blind phase I study of the safety, tolerability and immunogenicity of FLU-v no safety or tolerability concerns were identified at the doses administered (250 μg and 500 μg FLU-v) to the subjects in this clinical study and no safety or tolerability concerns were identified following administration of the adjuvant to the subjects (1). FLU-v vaccine candidate was demonstrated to be immunogenic in humans, as measured by ex vivo γ-interferon production (1).

Clinical experience with Montanide ISA 51 dates back to the 1990s and most trials were related to cancer and Acquired Immune Deficiency Syndrome (AIDS). Currently, cancer trials in melanoma, colorectal, prostate, cervical, brain cancer and leukemia are ongoing. Frequency of vaccination is often between 2 and 4 weeks, and the number of injections can reach up to 40. Route of immunization is most often subcutaneous and volume of injection can reach up to 3mL. Most common local reactions are local pain, tenderness, erythema and granuloma at the injection site. Less frequently, mild to moderate transient indurations and swelling are described. General reactions are mainly 'flu-like symptoms such as chills, fever and headaches. Lethargy and nausea are also observed. The intensity is usually mild or moderate. No biological changes are generally observed. As the Placebo vaccine is provided in a sealed single-use vial, overdose is highly unlikely (Influenza virus (FLU-v) vaccine Investigator's Brochure, Edition 2.0, 07 September 2015).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy non-pregnant females (as indicated by a negative blood pregnancy test done during the screening visit) between the ages of 18 and 60 years, inclusive;
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to one year) and men must agree to practice appropriate contraception (a combination of barrier and hormonal methods for women and a condom for men) from screening and until at least 30 days (up to Study Day 51 for females) and 90 days (up to Study Day 111 for males), after the last vaccination.
* A subject is in good health, as determined by a comprehensive clinical assessment {vital signs (heart rate, blood pressure, oral temperature)}, blood chemistry test (electrolytes, renal/kidney function, liver function, C-reactive protein, complete blood count), medical history, general physical examination, self-reported illness} and the clinical judgment of the investigator;
* Able to understand and comply with planned study procedures;
* Provides signed informed consent form

Exclusion Criteria:

* Has a known allergy to any of the components of the vaccine.
* Has a history of severe reaction following immunization.
* Persons with immune deficiency/disorder, whether due to genetic defect, immunodeficiency disease, or immunosuppressive therapy.
* Women who have a positive pregnancy test during the screening visit or who are breastfeeding.
* Has a history of any of the following (reported by subjects):

  * Acute disseminated encephalomyelitis (ADEM);
  * Neoplastic disease - current or previous;
  * Asthma or severe allergic disease;
  * Bleeding disorders
  * Chronic Hepatitis B and/or C infection;
  * Chronic liver disease;
  * Diabetes mellitus;
  * Guillain-Barré syndrome;
  * HIV;
  * Rheumatoid arthritis or other autoimmune diseases;
  * Severe renal disease;
  * Transplant recipients;
  * Unstable or progressive neurological disorders.
* Receipt of medicines/treatments that may affect evaluation of immunogenicity such as:

  * Oral or parenteral steroids, high-dose inhaled steroids (greater than 800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs (azathioprine (Imuran), cyclosporine (Neoral, Sandimmune, SangCya); monoclonal antibodies such as basiliximab (Simulect), daclizumab (Zinbryta), infliximab (Remicade), rituximab (MabThera), alemtuzumab (Campath and Lemtrada), omalizumab (Xolair), abatacept (Orencia), adalimumab (Humira and Exemptia) and etanercept (Enbrel)basiliximab (Simulect), daclizumab (Zenapax), and muromonab (Orthoclone OKT3); corticosteroids such as prednisone (Deltasone, Orasone); tacrolimus (Prograf, Advagraf, Protopic); Glatiramer acetate (Copaxone); Mycopehnolate (Cellcept); Sirolimus (Rapamune); (within 6 months of vaccination in this study)
  * Immunoglobulin or other blood products (plasma, blood cells, coagulation factors, haemoglobin)(within 3 months of vaccination in this study);
  * An experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month of vaccination in this study, or expects to receive an experimental agent (during the study period).
  * Influenza antiviral medication (Amantadine (Symmetrel); Rimantadine (Flumadine); Zanamivir (Relenza), Oseltamivir (Tamiflu) (within 4 weeks of vaccination in this study).
* Has received any influenza vaccine within 6 months of vaccination in this study.
* Has influenza-like illness (a sudden onset of symptoms and at least one of the four systemic symptoms-fever or feverishness, malaise, headache, myalgia and at least one of the three respiratory symptoms-cough, sore throat, shortness of breath) or acute respiratory infection (a sudden onset of symptoms and at least one of the four respiratory symptoms-cough, sore throat, shortness of breath, coryza (Rhinitis) and a clinician's judgement that the illness is due to an infection) within 6 months prior to vaccination in this study. These symptoms must have stopped the subject from carrying out their normal daily activities such as attending work or school for a period of at least 3 days.
* Has an acute illness, including an oral temperature greater than 38 degrees Celsius, within 1 week of vaccination.
* Has a history of alcohol or drug abuse within the last 2 years deemed unsuitable for inclusion by the investigator.
* Any abnormal haematology values and/or serum chemistries judged by the Investigator as clinically significant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Groeneveld, PhD, Principal Investigator — Isala
Locations (1):
- Isala, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Caparros-Wanderley W. Meta-Analysis and Potential Role of Preexisting Heterosubtypic Cellular Immunity Based on Variations in Disease Severity Outcomes for Influenza Live Viral Challenges in Humans. Clin Vaccine Immunol. 2015 Aug;22(8):949-56. doi: 10.1128/CVI.00101-15. Epub 2015 Jun 17. PMID 26084515
- [Background] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Mann A, Gilbert A, Balaratnam G, Wilkinson T, Lambkin-Williams R, Oxford J, Caparros-Wanderley W. A Synthetic Influenza Virus Vaccine Induces a Cellular Immune Response That Correlates with Reduction in Symptomatology and Virus Shedding in a Randomized Phase Ib Live-Virus Challenge in Humans. Clin Vaccine Immunol. 2015 Jul;22(7):828-35. doi: 10.1128/CVI.00098-15. Epub 2015 May 20. PMID 25994549
- [Background] Pleguezuelos O, Robinson S, Stoloff GA, Caparros-Wanderley W. Synthetic Influenza vaccine (FLU-v) stimulates cell mediated immunity in a double-blind, randomised, placebo-controlled Phase I trial. Vaccine. 2012 Jun 29;30(31):4655-60. doi: 10.1016/j.vaccine.2012.04.089. Epub 2012 May 8. PMID 22575166
- [Background] Stoloff GA, Caparros-Wanderley W. Synthetic multi-epitope peptides identified in silico induce protective immunity against multiple influenza serotypes. Eur J Immunol. 2007 Sep;37(9):2441-9. doi: 10.1002/eji.200737254. PMID 17668898
- [Background] van Doorn E, Pleguezuelos O, Liu H, Fernandez A, Bannister R, Stoloff G, Oftung F, Norley S, Huckriede A, Frijlink HW, Hak E. Evaluation of the immunogenicity and safety of different doses and formulations of a broad spectrum influenza vaccine (FLU-v) developed by SEEK: study protocol for a single-center, randomized, double-blind and placebo-controlled clinical phase IIb trial. BMC Infect Dis. 2017 Apr 4;17(1):241. doi: 10.1186/s12879-017-2341-9. PMID 28376743
- [Result] Pleguezuelos O, Dille J, de Groen S, Oftung F, Niesters HGM, Islam MA, Naess LM, Hungnes O, Aldarij N, Idema DL, Perez AF, James E, Frijlink HW, Stoloff G, Groeneveld P, Hak E. Immunogenicity, Safety, and Efficacy of a Standalone Universal Influenza Vaccine, FLU-v, in Healthy Adults: A Randomized Clinical Trial. Ann Intern Med. 2020 Apr 7;172(7):453-462. doi: 10.7326/M19-0735. Epub 2020 Mar 10. PMID 32150750
- See also: End of project reporting for the UNISEC Consortium — https://cordis.europa.eu/project/id/602012/reporting

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 195 subjects were screened. Of those, N=20 subjects were removed from the study prior randomisation due to:
  * lost to follow up n=3
  * didn't wish to continue after screening visit n=9
  * did not meet inclusion/exclusion criteria n=8
Groups:
- 2x Non-adjuvanted FLU-v: FLU-v on Day 0 and Day 21
  FLU-v: Subcutaneous injection in the upper arm with 500 ug of FLU-v as 0.5ml suspension in 0.01M HCl and 0.01M NaOH
- 1x Adjuvanted FLU-v: adjuvanted FLU-v on Day 0, saline (0.5mL) on Day 21
  adjuvanted FLU-v: Subcutaneous injection in the upper arm with 500ug of FLU-v emulsified in 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection
  Saline: Subcutaneous injection in the upper arm with 0.5ml of saline
- Non-adjuvanted Placebo: saline solution (0.5ml) on Day 0 and Day 21
  Saline: Subcutaneous injection in the upper arm with 0.5ml of saline
- Adjuvanted Placebo: Adjuvanted placebo on Day 0, saline (0.5mL) on Day 21
  Saline: Subcutaneous injection in the upper arm with 0.5ml of saline
  Adjuvanted placebo: Subcutaneous injection in the upper arm with an emulsion made with 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection
Period: Overall Study
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Started | 58 | 58 | 32 | 27
Completed | 58 | 50 | 32 | 24
Not Completed | 0 | 8 | 0 | 3
Not completed — Lost to Follow-up | 0 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A subject in 1x FLU-v adjuvanted group received 1x non-adjuvanted FLU-v. Subject completed the study but with this treatment, the subject could not be assigned to any group for analysis. This is the reason why 58 subjects were randomised to this group but only 57 were analysed, making the total subject number 174 rather than 175.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo | Total
Number analyzed (Participants) | 58 | 57 | 32 | 27 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.02 (13.691) | 40.12 (12.221) | 41.19 (12.458) | 39.07 (13.074) | 40.12 (12.806)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 30 | 18 | 13 | 97
  Male | 22 | 27 | 14 | 14 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 2
  Black of African descendant | 0 | 0 | 0 | 0 | 0
  White | 56 | 54 | 32 | 27 | 169
  Other | 1 | 2 | 0 | 0 | 3
  Unknown or not reported | 0 | 0 | 0 | 0 | 0
previous influenza vaccination [Count of Participants; unit: Participants] — Subjects were asked whether they had received previous influenza vaccinations and whether it was within 2 years or more from joining the trial. Population: This baseline measure was only analysed in the FAS population, that is the Full Analysis Set which includes all those subjects that completed vaccination and had at least pre-vaccination immunogenicity data and at least one post-vaccination time point.
  Participants
    Never received influenza vaccination | 37 | 29 | 15 | 18 | 99
    Received in the previous 2 years | 14 | 20 | 12 | 5 | 51
    Received over 2 years ago | 7 | 8 | 5 | 4 | 24
HAI titer at screening [Count of Participants; unit: Participants] — Serum samples were collected at screening (summer-autumn 2016) and later analysed for pre-existing neutralising antibodies against the main influenza strains that circulated in the Netherlands during the influenza season of 2016-2017 (B/Phuket/3073/2013, B/Brisbane/60/2008, A/Hong Kong/5738/2014 (H3N2) and A/Michigan/45/15 (H1N1)). The number of subjects with a HA titer for A strains ≥ 40 and with HA ≥ 80 for B strains was recorded in each group.
  Participants
    HAI≥80 B/Phuket/3073/2013 | 21 | 16 | 12 | 7 | 56
    HAI≥80 B/Brisbane/60/2008 | 18 | 19 | 12 | 7 | 56
    HAI≥40 A/Hong Kong/5738/2014 (H3N2) | 25 | 26 | 18 | 10 | 79
    HAI≥40 A/Michigan/45/15 (H1N1) | 23 | 29 | 16 | 11 | 79
    any of the above | 39 | 40 | 26 | 17 | 122

OUTCOME MEASURES:

1. Primary Outcome: CD4+ and CD8+ Th1 Cellular Immunogenicity on Day 42
Description: Comparison of the TH1 response in the treatment arms compared to placebo from baseline to day 42 following vaccination, calculated as the median fold change in the number of CD4+ and CD8+ T cells positive for IFN-gamma, TNF-alpha, IL-2 and CD107a. Fold change is calculated as the number of cells on day 42 divided by number of cells on day 0.
Time Frame: day 0 to day 42
Population: FAS population: Full Analysis Set corresponds to subjects that completed the vaccination successfully and provided samples for immunogenicity analysis for baseline (pre-vaccination) and at least one time point post-vaccination. Only samples with acceptable positive and negative controls were used in the analysis.
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
fold change
  IFN-gamma CD4+ | 0.5 [-0.2 to 1.1] | 5.9 [1.0 to 10.9] | 1.0 [-0.7 to 2.6] | 0.2 [-0.6 to 1.0]
  TNF-alpha CD4+ | 0.0 [-0.1 to 0.1] | 5.0 [-10.9 to 20.9] | 0.0 [-0.5 to 0.5] | 0.0 [-0.3 to 0.3]
  IL-2 CD4+ | 0.0 [-1.1 to 1.1] | 8.2 [-0.4 to 16.7] | 0.0 [-0.4 to 0.4] | 0.0 [-0.1 to 0.1]
  CD107a CD4+ | 0.0 [-0.4 to 0.4] | 2.0 [0.3 to 3.7] | 0.0 [-0.5 to 0.5] | 0.0 [-0.2 to 0.2]
  IFN-gamma CD8+ | 0.3 [-0.1 to 0.6] | 0.3 [-0.2 to 0.7] | 0.0 [-0.1 to 0.1] | 0.0 [-0.3 to 0.3]
  TNF-alpha CD8+ | 0.3 [0.0 to 0.6] | 0.3 [-0.6 to 1.3] | 0.0 [-0.6 to 0.6] | 0.0 [-0.1 to 0.1]
  IL-2 CD8+ | 0.5 [0.1 to 0.9] | 0.0 [-0.4 to 0.4] | 0.0 [-0.5 to 0.5] | 0.0 [-0.7 to 0.7]
  CD107a CD8+ | 0.0 [-0.2 to 0.2] | 0.0 [-0.5 to 0.5] | 0.0 [-0.2 to 0.2] | 0.0 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IFN-gamma from day 0 and to 42; Test type: Other — Inequality test; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — inequality test; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for TNF-alpha from day 0 to day 42; Test type: Other — inequality test; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Other — inequality test; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IL-2 from day 0 to day 42; Test type: Other — inequality test; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IL-2 from day 0 to day 42; Test type: Other — inequality test; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for CD107a from day 0 to day 42; Test type: Other — inequality test; p = 0.77, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for CD107a from day 0 to day 42; Test type: Other — inequality test; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for IFN-gamma from day 0 to day 42; Test type: Other — inequality test; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 1, analysis 9]; Test type: Other — inequality test; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for TNF-alpha from day 0 to day 42; Test type: Other — inequality test; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 1, analysis 11]; Test type: Other — inequality test; p = 0.156, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for IL-2 from day 0 to day 42; Test type: Other — inequality test; p = 0.125, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Test type: Other — inequality test; p = 0.89, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for CD107a from day 0 to day 42; Test type: Other — inequality test; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for CD107a from day 0 to day 42; Test type: Other — inequality test; p = 0.34, Wilcoxon (Mann-Whitney)

2. Primary Outcome: CD4+ and CD8+ Th1 Cellular Immunogenicity on Day 180
Description: Comparison of the TH1 response in the treatment arms compared to placebo from baseline to day 180 following vaccination, calculated as the median fold change in the number of CD4+ and CD8+ T cells positive for IFN-gamma, TNF-alpha, IL-2 and CD107a. Fold change is calculated as the number of cells on day 180 divided by number of cells on day 0.
Time Frame: Day 0 to day 180
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
fold change
  IFN-gamma CD4+ | 0.5 [0.2 to 1.2] | 4.4 [1.0 to 7.8] | 0.1 [-0.4 to 0.6] | 0.9 [-1.4 to 3.2]
  TNF-alpha CD4+ | 0.0 [0.0 to 0.0] | 0.6 [-3.5 to 4.8] | 0.0 [0.0 to 0.0] | 0.0 [-1.2 to 1.2]
  IL-2 CD4+ | 0.2 [-0.6 to 1.1] | 6.5 [2.1 to 10.9] | 0.0 [-0.2 to 0.2] | 0.0 [-0.1 to 0.1]
  CD107a CD4+ | 0.6 [-0.1 to 1.3] | 1.0 [0.2 to 1.8] | 0.0 [-0.1 to 0.1] | 0.6 [-0.7 to 1.9]
  IFN-gamma CD8+ | 0.0 [-0.5 to 0.6] | 0.2 [-0.4 to 0.7] | 0.0 [-0.6 to 0.6] | 0.0 [-0.5 to 0.5]
  TNF-alpha CD8+ | 0.1 [-0.5 to 0.6] | 0.2 [-0.2 to 0.6] | 0.1 [-0.7 to 0.9] | 0.1 [-1.8 to 1.85]
  IL-2 CD8+ | 0.3 [-0.3 to 0.7] | 0.0 [-0.6 to 0.6] | 0.0 [-0.3 to 0.3] | 0.0 [-0.4 to 0.4]
  CD107a CD8+ | 0.0 [-0.4 to 0.4] | 0.0 [-0.9 to 1.5] | 0.0 [-0.5 to 0.5] | 0.5 [-3.2 to 6.8]
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IFN-gamma from day 0 to day 180; Test type: Other — inequality test; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — inequality test; p = 0.030, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for TNF-alpha from day 0 to day 180; Test type: Other — inequality test; p = 0.87, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Other — inequality test; p = 0.075, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IL-2 from day 0 to day 180; Test type: Other — inequality test; p = 0.076, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for IL-2 from day 0 to day 180; Test type: Other — inequality test; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD4+ T cells positive for CD107a from day 0 to day 180; Test type: Other — inequality test; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Other — inequality test; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for IFN-gamma from day 0 to day 180; Test type: Other — inequality test; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Other — inequality test; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for TNF-alpha from day 0 to day 180; Test type: Other — inequality; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Other — inequality test; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for IL2 from day 0 to day 180; Test type: Other — inequality test; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for IL2 from day 0 to day 180; Test type: Other — inequality test; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the difference in median fold increase in number of CD8+ T cells positive for CD107a from day 0 to day 180; Test type: Other — inequality test; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 2, analysis 15]; Test type: Other — inequality; p = 0.23, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Percentage of TH1 Cytokine Responders (Responders Defined as Those With >2 Fold Median Increase From Baseline in CD4+ and CD8+ T-cells Positive for Particular Cytokine)
Description: To compare the number of subjects that showed at least a two-fold increase on day 42 and day 180 following vaccination in the number of CD4+and CD8+ T-cells secreting TH1 cytokines in all groups.
Time Frame: prevaccination, day 42 (21 days after last vaccination) and day 180.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
Participants
  IFNg+CD4+ day 42: number analyzed (Participants) | 51 | 44 | 27 | 19
  IFNg+CD4+ day 42 | 23 | 40 | 13 | 8
  TNFalpha+ CD4+ day 42: number analyzed (Participants) | 52 | 44 | 27 | 18
  TNFalpha+ CD4+ day 42 | 16 | 33 | 12 | 9
  IL2+ CD4+ day 42: number analyzed (Participants) | 52 | 44 | 27 | 19
  IL2+ CD4+ day 42 | 23 | 36 | 13 | 4
  CD107a+ CD4+ day 42: number analyzed (Participants) | 47 | 38 | 23 | 14
  CD107a+ CD4+ day 42 | 22 | 26 | 8 | 4
  IFNg+ CD4+ day 180: number analyzed (Participants) | 53 | 44 | 27 | 19
  IFNg+ CD4+ day 180 | 26 | 37 | 8 | 11
  TNFa+ CD4+ day 180: number analyzed (Participants) | 53 | 44 | 27 | 19
  TNFa+ CD4+ day 180 | 17 | 26 | 9 | 9
  IL-2+ CD4+ day 180: number analyzed (Participants) | 53 | 44 | 27 | 19
  IL-2+ CD4+ day 180 | 26 | 39 | 13 | 9
  CD107a+ CD4+ day 180: number analyzed (Participants) | 50 | 37 | 22 | 14
  CD107a+ CD4+ day 180 | 24 | 21 | 5 | 8
  IFN-gamma day 42 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 18
  IFN-gamma day 42 CD8+ | 22 | 16 | 9 | 4
  TNF-alpha day 42 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 18
  TNF-alpha day 42 CD8+ | 22 | 23 | 10 | 6
  IL2 day 42 CD8+: number analyzed (Participants) | 52 | 44 | 27 | 19
  IL2 day 42 CD8+ | 25 | 17 | 9 | 8
  CD107a day 42 CD8+: number analyzed (Participants) | 47 | 44 | 27 | 18
  CD107a day 42 CD8+ | 23 | 19 | 5 | 2
  IFN-gamma day 180 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 19
  IFN-gamma day 180 CD8+ | 27 | 22 | 13 | 7
  TNF-alpha day 180 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 19
  TNF-alpha day 180 CD8+ | 21 | 18 | 14 | 12
  IL2 day 180 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 19
  IL2 day 180 CD8+ | 11 | 16 | 8 | 5
  CD107a day 180 CD8+: number analyzed (Participants) | 53 | 44 | 27 | 19
  CD107a day 180 CD8+ | 19 | 24 | 8 | 8
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ IFNgamma responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.80, Chi-squared
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ IFNgamma responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ TNF alpha responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.23, Chi-squared
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ TNF alpha responders on day 42. Differences considered significant if p-value <0.05; Test type: Other; p = 0.056, Chi-squared
Statistical Analysis 5: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ IL-2 responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.74, Chi-squared
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ IL-2 responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 7: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ CD107a responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.34, Fisher Exact
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ CD107a responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.010, Fisher Exact
Statistical Analysis 9: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ IFNgamma responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.096, Chi-squared
Statistical Analysis 10: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ IFNgamma responders on day 180.Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.049, Fisher Exact
Statistical Analysis 11: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ TNF alpha responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.91, Chi-squared
Statistical Analysis 12: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ TNF alpha responders on day 180. Differences considered significant if p-value <0.05; Test type: Other; p = 0.39, Chi-squared
Statistical Analysis 13: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ IL-2 responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.94, Chi-squared
Statistical Analysis 14: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ IL-2 responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p < 0.001, Fisher Exact
Statistical Analysis 15: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD4+ CD107a responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.044, Fisher Exact
Statistical Analysis 16: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD4+ CD107a responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.98, Fisher Exact
Statistical Analysis 17: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ IFN-gamma responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.48, Chi squared or Fisher's exact test
Statistical Analysis 18: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ IFN-gamma responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.28, Chi squared or Fisher's exact test
Statistical Analysis 19: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ TNF-alpha responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.70, Chi squared or Fisher's exact test
Statistical Analysis 20: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ TNF-alpha responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.175, Chi squared or Fisher's exact test
Statistical Analysis 21: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ IL2 responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.24, Chi squared or Fisher's exact test
Statistical Analysis 22: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ IL2 responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.80, Chi squared or Fisher's exact test
Statistical Analysis 23: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ CD107a responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.023, Chi squared or Fisher's exact test
Statistical Analysis 24: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ CD107a responders on day 42. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.015, Chi squared or Fisher's exact test
Statistical Analysis 25: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ IFN-gamma responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.81, Chi squared or Fisher's exact test
Statistical Analysis 26: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ IFN-gamma responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.34, Chi squared or Fisher's exact test
Statistical Analysis 27: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ TNF-alpha responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.30, Chi squared or Fisher's exact test
Statistical Analysis 28: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ TNF-alpha responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.105, Chi squared or Fisher's exact test
Statistical Analysis 29: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ IL2 responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.38, Chi squared or Fisher's exact test
Statistical Analysis 30: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ IL2 responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.44, Chi squared or Fisher's exact test
Statistical Analysis 31: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of CD8+ CD107a responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.58, Chi squared or Fisher's exact test
Statistical Analysis 32: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of CD8+ CD107a responders on day 180. Differences considered significant if p-value <0.05; Test type: Other — inequality test; p = 0.43, Chi squared or Fisher's exact test

4. Primary Outcome: Percentage of CD4+ and CD8+ TH1 Cytokine Responders Determined by Mixture Models for Single-cell Assays (MIMOSA)
Description: To compare the number of subjects identified as responders for cytokine markers as determined by MIMOSA analysis (Responders based on a false discovery rate derived P-value <0.05).
Time Frame: day 0 to day 42 and day 180
Population: FAS: Full Analysis Set corresponds to subjects that completed the vaccination successfully and provided samples for immunogenicity analysis for baseline (pre-vaccination) and at least one time point post-vaccination. Only samples with acceptable positive and negative controls were used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
Participants
  IFN-gamma day 42 CD4+: number analyzed (Participants) | 54 | 50 | 30 | 23
  IFN-gamma day 42 CD4+ | 7 | 38 | 1 | 2
  TNF-alpha day 42 CD4+: number analyzed (Participants) | 55 | 50 | 30 | 22
  TNF-alpha day 42 CD4+ | 3 | 22 | 1 | 0
  IL-2 day 42 CD4+: number analyzed (Participants) | 55 | 50 | 30 | 23
  IL-2 day 42 CD4+ | 1 | 28 | 1 | 0
  CD107a day 42 CD4+: number analyzed (Participants) | 51 | 48 | 29 | 21
  CD107a day 42 CD4+ | 1 | 5 | 1 | 0
  IFN-gamma day 180 CD4+: number analyzed (Participants) | 56 | 49 | 30 | 21
  IFN-gamma day 180 CD4+ | 8 | 31 | 2 | 1
  TNF-alpha day 180 CD4+: number analyzed (Participants) | 56 | 49 | 30 | 21
  TNF-alpha day 180 CD4+ | 2 | 12 | 1 | 0
  IL-2 day 180 CD4+: number analyzed (Participants) | 56 | 49 | 30 | 21
  IL-2 day 180 CD4+ | 1 | 28 | 1 | 0
  CD107a day 180 CD4+: number analyzed (Participants) | 53 | 44 | 25 | 19
  CD107a day 180 CD4+ | 2 | 4 | 2 | 1
  IFN-gamma day 42 CD8+: number analyzed (Participants) | 56 | 50 | 30 | 22
  IFN-gamma day 42 CD8+ | 3 | 3 | 0 | 0
  TNF-alpha day 42 CD8+: number analyzed (Participants) | 56 | 50 | 30 | 22
  TNF-alpha day 42 CD8+ | 0 | 1 | 0 | 0
  IL2 day 42 CD8+: number analyzed (Participants) | 56 | 50 | 30 | 23
  IL2 day 42 CD8+ | 0 | 0 | 0 | 0
  CD107a day 42 CD8+: number analyzed (Participants) | 55 | 50 | 30 | 22
  CD107a day 42 CD8+ | 0 | 0 | 0 | 0
  IFN-gamma day 180 CD8+: number analyzed (Participants) | 56 | 49 | 30 | 21
  IFN-gamma day 180 CD8+ | 4 | 3 | 0 | 1
  TNF-alpha day 180 CD8+: number analyzed (Participants) | 56 | 49 | 30 | 21
  TNF-alpha day 180 CD8+ | 1 | 1 | 0 | 0
  IL2 day 180 CD8+: number analyzed (Participants) | 56 | 49 | 30 | 21
  IL2 day 180 CD8+ | 0 | 0 | 0 | 0
  CD107a day 180 CD8+: number analyzed (Participants) | 56 | 49 | 30 | 21
  CD107a day 180 CD8+ | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IFN-gamma at day 42; Test type: Other — inequality test; p = 0.25, Fisher Exact
Statistical Analysis 2: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing TNF-alpha at day 42; Test type: Other — inequality test; p = 1.0, Fisher Exact
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IL-2 at day 42; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 4: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing CD107a at day 42; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 5: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IFN-gamma at day 42; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing TNF-alpha at day 42; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 7: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IL2 at day 42; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing CD107a at day 42; Test type: Other — inequality test; p = 0.31, Fisher Exact
Statistical Analysis 9: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IFN-gamma at day 180; Test type: Other — inequality test; p = 0.48, Fisher Exact
Statistical Analysis 10: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing TNF-alpha at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 11: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IL2 at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 12: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing CD107a at day 180; Test type: Other — inequality test; p = 0.59, Fisher Exact
Statistical Analysis 13: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IFN-gamma at day 180; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 14: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing TNF-alpha at day 180; Test type: Other — inequality test; p = 0.013, Fisher Exact
Statistical Analysis 15: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing IL2 at day 180; Test type: Other — inequality; p < 0.001, Chi-squared
Statistical Analysis 16: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD4+ T-cell producing CD107a at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 17: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing IFN-gamma at day 42; Test type: Other — inequality test; p = 0.55, Fisher Exact
Statistical Analysis 18: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing IFN-gamma at day 42; Test type: Other — inequality test; p = 0.55, Fisher Exact
Statistical Analysis 19: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing TNF-alpha at day 42; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 20: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing IFN-gamma at day 180; Test type: Other — inequality test; p = 0.29, Fisher Exact
Statistical Analysis 21: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing TNF-alpha at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 22: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing IFN-gamma at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 23: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing TNF-alpha at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact
Statistical Analysis 24: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of responders determined by MIMOSA analysis of CD8+ T-cell producing CD107a at day 180; Test type: Other — inequality test; p = 1.00, Fisher Exact

5. Primary Outcome: IFN-gamma Responses Measured by ELISA
Description: Median fold change in IFN-gamma secretion from PBMCs stimulated in vitro with FLU-v antigens. IFN-gamma secretion was measured by ELISA.Fold change was measured as secretion on day 42 divided by secretion on day 0, and secretion on day 180 divided by secretion on day 0.
Time Frame: day 0 to day 42, day 0 to day 180
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
fold change
  Day 42: number analyzed (Participants) | 47 | 43 | 25 | 20
  Day 42 | 0.8 [-2.3 to 3.9] | 59.0 [33.3 to 84.7] | 1.0 [-0.8 to 2.8] | 1.0 [-2.4 to 4.4]
  Day 180: number analyzed (Participants) | 48 | 43 | 23 | 20
  Day 180 | 1.0 [0.7 to 1.3] | 27.3 [5.2 to 49.4] | 1.0 [-1.4 to 3.4] | 0.9 [-0.0 to 1.9]
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of median fold-increase in IFN-gamma secretion as measured by ELISA on day 42. p<0.05 considered statistically significant; Test type: Other — inequality test; p = 0.59, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other — inequality test; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of median fold-increase in IFN-gamma secretion as measured by ELISA on day 180. p<0.05 considered statistically significant; Test type: Other — inequality test; p = 0.61, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Other — inequality test; p < 0.001, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Percentage of Responders on Day 42 and Day 180 for IFNgamma Secretion by PBMCs
Description: Responders were defined as subjects having at least a two-fold increase in the amount of IFNg secreted on day 42 and day 180 compared the amount secreted on day 0. IFNg was measured by ELISA
Time Frame: prevaccination (day 0) to postvaccination (day 42 and day 180)
Population: FAS: Full Analysis Set including subjects that completed vaccination and provided immunogenicity samples for prevaccination and at least one post-vaccination time point (day 42 or day 180). Only samples that meet the acceptance criteria based on the positive and negative controls were used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
Participants
  day 42: number analyzed (Participants) | 47 | 44 | 25 | 20
  day 42 | 28 | 42 | 10 | 9
  day 180: number analyzed (Participants) | 48 | 43 | 23 | 20
  day 180 | 22 | 40 | 13 | 11
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of number of responders on day 42. A subject was considered a "responder" if an increase of secreted IFNgamma of at least two fold was observed from day 0 to day 42; Test type: Other; p = 0.113, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of number of responders on day 180. A subject was considered a "responder" if an increase of secreted IFNgamma of at least two fold was observed from day 0 to day 180; Test type: Other; p = 0.399, Chi-squared
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Other; p < 0.001, Fisher Exact

7. Primary Outcome: Solicited AEs
Description: To evaluate the solicited AEs in all subjects
Time Frame: until 21 days after the last dosing of the study vaccine
Population: Safety Population: All subjects that received at least one vaccination
Measure: Number; unit: Events
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 57 | 32 | 27
Events
  All solicited AEs | 275 | 485 | 149 | 147
  Solicited AEs unrelated to vaccination | 12 | 13 | 8 | 0
  Solicited AEs unlikely related to vaccination | 72 | 74 | 71 | 34
  Solicited AEs possibly related to vaccination | 108 | 134 | 64 | 39
  Solicited AEs probably related to vaccination | 16 | 16 | 0 | 12
  Solicited AEs definately related to vaccination | 67 | 248 | 6 | 62
  Mild solicited AEs | 210 | 339 | 124 | 111
  Moderate solicited AEs | 59 | 132 | 24 | 34
  Severe solicited AEs | 6 | 14 | 1 | 2

8. Secondary Outcome: Antibody Responses to FLU-v
Description: To evaluate the IgG levels as a measure of antibody responses to FLU-v on day 0 (baseline) and on days 42 and 180 following FLU-v vaccination. IgG antibodies were measured by ELISA. The geometric mean for each treatment group was provided.
Time Frame: prevaccination, day 42 (21 days after last vaccination) and day 180.
Population: FAS: Full Analysis Set includes all subjects that completed the vaccination successfully and provided samples for immunogenicity analysis at baseline (Pre-vaccination) and at least one time point post-vaccination.
Measure: Geometric Mean (Standard Error); unit: IgG ng/ml
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
IgG ng/ml
  day 0 | 499.11 (103.19) | 362.86 (82.93) | 331.16 (59.00) | 371.89 (67.47)
  day 42 | 2593.02 (1652.34) | 8740.48 (2432.90) | 336.37 (58.92) | 381.17 (61.18)
  day 180 | 1276.34 (344.52) | 4769.16 (1131.67) | 344.88 (66.57) | 387.26 (61.48)
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of geometric mean IgG titers specific to FLU-v antigens on day 42 post-vaccination; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of geometric mean IgG titers specific to FLU-v antigens on day 42; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of geometric mean IgG titers specific to FLU-v antigens on day 180; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of geometric mean IgG titers specific to FLU-v antigens on day 180; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Th2 Cytokine Responses (IL-4)
Description: To evaluate the level of TH2 cytokines (IL-4) from baseline in all groups 42 and 180 days following FLU-v vaccination.
Time Frame: prevaccination, day 42 (21 days after last vaccination) and day 180.
Population: FAS: Full Analysis Set includes all subjects that completed the vaccination successfully and provided samples for immunogenicity analysis at baseline (Pre-vaccination) and at least one time point post-vaccination. Only samples that met the acceptance criteria based on positive and negative controls were used in the analysis
Measure: Number; unit: percentage of responders
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
percentage of responders
  IL-4+CD4+ cells day 42 | NA — Below level of detection | NA — below level of detection | NA — below level of detection | NA — below level of detection
  IL-4+ CD8+ cells day 42 | NA — below level of detection | NA — below level of detection | NA — below level of detection | NA — below level of detection
  IL-4+ CD4+ cells day 180 | NA — below level of detection | NA — below level of detection | NA — below level of detection | NA — below level of detection
  IL-4+ CD8+ cells day 180 | NA — below level of detection | NA — below level of detection | NA — below level of detection | NA — below level of detection

10. Other Pre Specified Outcome: Unsolicited AEs and SAEs
Description: To evaluate unsolicited AEs and SAEs in all subjects
Time Frame: From the start of the vacciantion until study completion for each subject, approximately no more than 7 months
Population: Safety Population: all subjects that received at least one vaccination
Measure: Number; unit: events
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 57 | 32 | 27
events
  All unsolicited AEs | 19 | 24 | 13 | 9
  Unsolicited AEs unrelated to the vaccine | 8 | 11 | 5 | 5
  Unsolicited AEs unlikely related to the vacccine | 4 | 8 | 7 | 3
  Unsolicited AEs possibly related to the vacccine | 5 | 4 | 1 | 1
  Unsolicited AEs probably related to the vaccine | 0 | 0 | 0 | 0
  Unsolicited AEs definately related to the vaccine | 2 | 1 | 0 | 0
  Mild unsolicited AEs | 15 | 16 | 10 | 4
  Moderate unsolicited AEs | 3 | 4 | 1 | 5
  Severe unsolicited AEs | 1 | 3 | 2 | 0
  Severe Adverse Events | 2 | 3 | 0 | 0

11. Other Pre Specified Outcome: Percentage of Participants Who Tested Positive for Influenza Strains
Description: During the influenza season (Dec 2016 to March 2017), fully vaccinated subjects will contact the trial center immediately if they feel unwell for 24h, with a sudden onset of flu-like symptoms. The medical staff will arrange for a nasopharyngeal swab to be performed if the subject has at least one respiratory (cough, sore throat, shortness of breath, runny nose, stuffy nose, sneezing and earache) and one systemic symptom (fever, malaise, headache and myalgia (muscle and joint pain). Swabs should be taken from the reported subjects within 3 days from the trial center being contacted or within 4 days of the onset of symptoms, whatever time is shorter.
Time Frame: For up to 4 months during the influenza season
Population: FAS: Full Analysis Set includes subjects that completed vaccination and provided samples to measure immunogenicity data prevaccination (day 0) and at least one time point post vaccination (day 42 or day 180)
Measure: Number; unit: percentage of subjects
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
percentage of subjects
  positive for influenza A strains | 5.2 | 7.8 | 6.3 | 19.2
  positive for influenza B strains | 0.0 | 2.0 | 3.1 | 3.8
  positive for influenza H1 strains | 0.0 | 0.0 | 0.0 | 0.0
  positive for influenza H3 strains | 5.2 | 7.8 | 6.3 | 19.2
  positive for any influenza strain | 5.2 | 9.8 | 9.4 | 23.1
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Differences in the infection rates against any of the strains tested between treatment group and corresponding placebo; Test type: Other; p = 0.662, Fisher Exact
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Differences in the infection rates against any of the strains tested between treatment group and corresponding placebo; Test type: Other; p = 0.168, Fisher Exact

12. Other Pre Specified Outcome: Severity of Symptoms in RT-PCR Influenza-confirmed Subjects.
Description: Subjects recorded daily influenza symptoms from December 2016 up to March 2017. Subjects with a sudden onset of at least one respiratory and one systemic symptom were swabbed. If the results were positive for influenza then the symptoms were included in the analysis. The duration of symptoms was recorded as the number of symptomatic days during the influenza episode. Fever (≥38oC), malaise, headache, myalgia (muscle and joint pain), cough, sore throat, shortness of breath, runny nose, stuffy nose, sneezing and earache were scored on a severity scale of 0 to 3 (0: no symptom, 1: mild, 2: moderate, 3: severe). The daily severity score was the sum of the severity score for all symptoms listed above on a single day. The total score was the sum of all daily scores during the influenza episode. The peak score was the highest daily score during the influenza episode. The average score was the total score divided by the number of days the influenza episode lasted.
Time Frame: Symptoms experienced during an influenza infection episode, approximately 7-10 days.
Population: FAS: Full Analysis Set includes subjects that completed vaccination and provided samples to assess immunogenicity at pre-vaccination (day 0) and at least one post-vaccination time point (day 42 or day 180).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
units on a scale
  total symptom score | 113.67 (50.87) | 30.80 (8.46) | 57.33 (13.28) | 55.17 (12.96)
  total symptom peak | 17.67 (3.48) | 13.80 (1.16) | 15.33 (1.20) | 16.50 (2.73)
  average severity symptom score | 10.63 (1.13) | 10.92 (1.61) | 8.59 (1.44) | 13.76 (2.12)
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney); The study was not powered to detected statistical significant differences in this outcome
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney); Study not powered to detect statistically significant differences

13. Other Pre Specified Outcome: Duration of Influenza Symptoms in RT-PCR Confirmed Infected Subjects.
Description: Subjects recorded daily influenza symptoms from December 2016 up to March 2017. Subjects with a sudden onset of at least one respiratory and one systemic symptom were swabbed. If the results were positive for influenza then the symptoms were included in the analysis. The duration of symptoms was recorded as the number of symptomatic days during the influenza episode. The following symptoms were recorded: fever (≥38oC), malaise, headache, myalgia (muscle and joint pain), cough, sore throat, shortness of breath, runny nose, stuffy nose, sneezing and earache.
Time Frame: During an influenza episode
Population: FAS population: subjects that completed the vaccination and had immunogenicity data at pre-vaccination and at least one time point post-vaccination.
Measure: Mean (Standard Error); unit: days
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
Number analyzed (Participants) | 58 | 51 | 32 | 26
days | 11.67 (5.61) | 3.20 (1.07) | 7.33 (2.19) | 4.00 (0.86)
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison in the duration of symptoms between treatment group and corresponding placebo; Test type: Other; p = 0.513, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the duration of symptoms between treatment group and corresponding placebo; Test type: Other; p = 0.578, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of total symptom score between treatment group and corresponding placebo; Test type: Other; p = 0.513, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the total symptom score between treatment group and corresponding placebo; Test type: Other; p = 0.200, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the symptom peak between treatment group and corresponding placebo; Test type: Other; p = 0.658, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the symptom peak between treatment group and corresponding placebo; Test type: Other; p = 0.640, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: 2x Non-adjuvanted FLU-v vs Non-adjuvanted Placebo; Comparison of the average symptom score between treatment group and corresponding placebo; Test type: Other; p = 0.127, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v vs Adjuvanted Placebo; Comparison of the average symptom score between treatment group and corresponding placebo; Test type: Other; p = 0.201, Wilcoxon (Mann-Whitney)

14. Post Hoc Outcome: Effect of Influenza Vaccination in Previous 2 Years on Immunogenicity
Description: Antigen specific responders in FLU-v vaccinated arms compared to combined placebo group, grouped into those who had recieved an influenza vaccination within the previous 2 years and those who had not ever received a previous influenza vaccination. Responders were defined as those having a ≥2-fold increase in response in IFN-gamma secretion by peripheral blood mononuclear cells from day 0 to day 42 or day 180, as measured by enzyme-linked immunosorbent assay. The combined placebo group includes participants randomly assigned to adjuvanted placebo and those assigned to nonadjuvanted placebo.
Time Frame: day 0 to day 42, day 0 to day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- 2x Non-adjuvanted FLU-v, Previous Vaccination Within 2 Years: participants who had received an influenza vaccination in the previous 2 years, and who received FLU-v on Day 0 and Day 21 FLU-v: Subcutaneous injection in the upper arm with 500 ug of FLU-v as 0.5ml suspension in 0.01M HCl and 0.01M NaOH
- 1x Adjuvanted FLU-v, Previous Vaccination Within 2 Years: participants who had received an influenza vaccination in the previous 2 years, and who received adjuvanted FLU-v on Day 0, saline (0.5mL) on Day 21
  adjuvanted FLU-v: Subcutaneous injection in the upper arm with 500ug of FLU-v emulsified in 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection Saline: Subcutaneous injection in the upper arm with 0.5ml of saline
- Combined Placebo, Previous Vaccination Within 2 Years: participants who had received an influenza vaccination in the previous 2 years, and who received either non-adjuvanted placebo or adjuvanted placebo
  Non-adjuvanted Placebo: saline solution (0.5ml) on Day 0 and Day 21
  Adjuvanted Placebo: Adjuvanted placebo on Day 0, saline (0.5mL) on Day 21
  Saline: Subcutaneous injection in the upper arm with 0.5ml of saline Adjuvanted placebo: Subcutaneous injection in the upper arm with an emulsion made with 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection
- 2x Non-adjuvanted FLU-v, no Previous Vaccination: Participants who had not ever previously received an influenza vaccination, and who received FLU-v on Day 0 and Day 21
  FLU-v: Subcutaneous injection in the upper arm with 500 ug of FLU-v as 0.5ml suspension in 0.01M HCl and 0.01M NaOH
- 1x Adjuvanted FLU-v, no Previous Vaccination: participants who had not ever previously received an influenza vaccination, and who received adjuvanted FLU-v on Day 0, saline (0.5mL) on Day 21
  adjuvanted FLU-v: Subcutaneous injection in the upper arm with 500ug of FLU-v emulsified in 0.25ml of Montanide ISA-51 adjuvant (Seppic, France) and 0.25ml of water for injection Saline: Subcutaneous injection in the upper arm with 0.5ml of saline
- Combined Placebo, no Previous Vaccination: participants who had not ever previously received an influenza vaccination, and who received either non-adjuvanted placebo or adjuvanted placebo
  Non-adjuvanted Placebo: saline solution (0.5ml) on Day 0 and Day 21
  Adjuvanted Placebo: Adjuvanted placebo on Day 0, saline (0.5mL) on Day 21
Arm/Group | 2x Non-adjuvanted FLU-v, Previous Vaccination Within 2 Years | 1x Adjuvanted FLU-v, Previous Vaccination Within 2 Years | Combined Placebo, Previous Vaccination Within 2 Years | 2x Non-adjuvanted FLU-v, no Previous Vaccination | 1x Adjuvanted FLU-v, no Previous Vaccination | Combined Placebo, no Previous Vaccination
Number analyzed (Participants) | 14 | 18 | 16 | 37 | 25 | 33
Participants
  Responders on day 42: number analyzed (Participants) | 12 | 15 | 13 | 31 | 21 | 24
  Responders on day 42 | 6 | 13 | 6 | 20 | 21 | 10
  Responders on day 180: number analyzed (Participants) | 10 | 15 | 13 | 33 | 21 | 25
  Responders on day 180 | 5 | 13 | 8 | 15 | 21 | 15
Statistical Analysis 1: Comparison: 2x Non-adjuvanted FLU-v, Previous Vaccination Within 2 Years vs Combined Placebo, Previous Vaccination Within 2 Years; comparison between groups on day 42; Test type: Other — inequality test; p = 0.85, Chi-squared
Statistical Analysis 2: Comparison: 1x Adjuvanted FLU-v, Previous Vaccination Within 2 Years vs Combined Placebo, Previous Vaccination Within 2 Years; comparison between groups on day 42; Test type: Other — inequality test; p = 0.042, Fisher Exact
Statistical Analysis 3: Comparison: 2x Non-adjuvanted FLU-v, Previous Vaccination Within 2 Years vs Combined Placebo, Previous Vaccination Within 2 Years; comparison between groups on day 180; Test type: Other — inequality test; p = 0.69, Fisher Exact
Statistical Analysis 4: Comparison: 1x Adjuvanted FLU-v, Previous Vaccination Within 2 Years vs Combined Placebo, Previous Vaccination Within 2 Years; comparison between groups on day 180; Test type: Other — inequality test; p = 0.198, Fisher Exact
Statistical Analysis 5: Comparison: 2x Non-adjuvanted FLU-v, no Previous Vaccination vs Combined Placebo, no Previous Vaccination; comparison between groups on day 42; Test type: Other — inequality test; p = 0.092, Chi-squared
Statistical Analysis 6: Comparison: 1x Adjuvanted FLU-v, no Previous Vaccination vs Combined Placebo, no Previous Vaccination; comparison of groups on day 42; Test type: Other — inequality test; p < 0.001, Chi-squared
Statistical Analysis 7: Comparison: 2x Non-adjuvanted FLU-v, no Previous Vaccination vs Combined Placebo, no Previous Vaccination; comparison of groups on day 180; Test type: Other — inequality test; p = 0.27, Chi-squared
Statistical Analysis 8: Comparison: 1x Adjuvanted FLU-v, no Previous Vaccination vs Combined Placebo, no Previous Vaccination; comparisons between groups on day 180; Test type: Other — inequality test; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: From vaccination to study completion (approx. 7 months)
Description: Solicited Adverse Events were collected for 21 days after each vaccination. Subjects had to fill in the AEs diary card daily and return to the clinic on the next scheduled visit.
  Unsolicited Adverse Events and Severe Adverse Events were collected at any time during the study directly to the PI or study doctor.
Arm/Group | 2x Non-adjuvanted FLU-v | 1x Adjuvanted FLU-v | Non-adjuvanted Placebo | Adjuvanted Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57 | 0/32 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/58 | 2/57 | 0/32 | 0/27
Other Adverse Events (participants affected / at risk) | 41/58 | 50/57 | 27/32 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2x Non-adjuvanted FLU-v (N=58) | 1x Adjuvanted FLU-v (N=57) | Non-adjuvanted Placebo (N=32) | Adjuvanted Placebo (N=27)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol problem (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2x Non-adjuvanted FLU-v (N=58) | 1x Adjuvanted FLU-v (N=57) | Non-adjuvanted Placebo (N=32) | Adjuvanted Placebo (N=27)
Lymphadenopathy (Blood and lymphatic system disorders) | 7 (8) | 4 (4) | 3 (4) | 4 (4)
diarrhoea (Gastrointestinal disorders) | 6 (8) | 8 (9) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6) | 2 (2) | 0 (0)
Fatigue (General disorders) | 14 (16) | 17 (25) | 11 (12) | 6 (6)
Influenza like illness (General disorders) | 11 (12) | 18 (19) | 10 (11) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 14 (15) | 13 (14) | 6 (6)
Decreased apetite (Metabolism and nutrition disorders) | 1 (1) | 11 (12) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (7) | 6 (7) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (12) | 6 (6) | 4 (5)
Headache (Nervous system disorders) | 13 (20) | 19 (30) | 14 (18) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 17 (20) | 8 (9) | 3 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 11 (12) | 9 (12) | 8 (9)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 15 (19) | 14 (17) | 7 (8)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 17 (19) | 14 (20) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (8) | 1 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 13 (15) | 38 (40) | 0 (0) | 6 (6)
Injection site pain (General disorders) | 4 (6) | 39 (46) | 4 (4) | 11 (12)
Injection site swelling (General disorders) | 6 (7) | 38 (39) | 0 (0) | 7 (7)
Injection site warmth (General disorders) | 7 (9) | 29 (30) | 1 (1) | 6 (7)
Injection site pruritus (General disorders) | 9 (10) | 22 (23) | 0 (0) | 10 (14)
Injection site induration (General disorders) | 16 (18) | 49 (49) | 0 (0) | 10 (11)
Haematoma at Injection Site (General disorders) | 5 (6) | 19 (19) | 0 (0) | 5 (5)
Herpes simplex (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment stopped early at 175 subjects instead of 222. Dropout rate was lower than anticipated (4% vs 20%). The number of participants recruited was considered to be sufficient to provide statistically significant data in the primary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02962908/ICF_000.pdf
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02962908/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT02962908/SAP_002.pdf